CLINICAL TRIAL: NCT03215264
Title: Phase I/II Trial of Regorafenib, Hydroxychloroquine, and Entinostat in Metastatic Colorectal Cancer
Brief Title: To Determine the Safety of Regorafenib, Hydroxychloroquine, and Entinostat Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 31216
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Hydroxychloroquine; entinostat; regorafenib

STUDY DESIGN:
Intervention Model Description: Standard 3+3 design to determine the maximum tolerated dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose level 1 (Experimental): Regorafenib 160mg daily 1-21 of 28-day cycle , Entinostat 3mg weekly, HCQ 600mg daily.
  Interventions: Drug: hydroxychloroquine; Drug: entinostat; Drug: regorafenib
- Dose level 2 (Experimental): Regorafenib 160mg daily 1-21 of 28-day cycle Entinostat 5mg weekly, HCQ 600mg daily
  Interventions: Drug: hydroxychloroquine; Drug: entinostat; Drug: regorafenib
- Dose level 3 (Experimental): Regorafenib 160mg daily 1-21 of 28-day cycle, Entinostat 5mg weekly, HCQ 600mg BID (1200mg daily).
  Interventions: Drug: hydroxychloroquine; Drug: entinostat; Drug: regorafenib

INTERVENTIONS:
Drug: hydroxychloroquine — 600-1200mg daily
  Other Names: Plaquenil · Quineprox
Drug: entinostat — 3-5mg weekly
  Other Names: DB11841
Drug: regorafenib — 160mg daily
  Other Names: Stivarga

SUMMARY:
The main purpose of this study is to find the best dose of hydroxychloroquine (HCQ) when given in combination with regorafenib and entinostat.

DETAILED DESCRIPTION:
This was a 3+3 phase I trial of HCQ and entinostat with regorafenib in patients with metastatic CRC. The primary objective was safety and the secondary objective was clinical efficacy. The trial was intended to be a Phase 1/2 trial, but the trial never moved forward to Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of metastatic colorectal cancer
* Measurable disease based on modified RECIST 1.1 criteria
* Patients should have received adequate therapy with prior 5-fluorouracil, oxaliplatin, and irinotecan, unless contra-indicated, not tolerated or declined.
* No prior therapy with regorafenib or other anti-angiogenic tyrosine kinase inhibitor
* No prior or current therapy with an HDAC inhibitor
* Age 18 years or older
* ECOG performance status of 0 or 1
* If a female of childbearing potential, has a negative serum blood pregnancy test during screening and a negative urine pregnancy test within 3 days prior to receiving the first dose of study drug. If the screening serum test is done within 3 days prior to receiving the first dose of study drug, a urine test is not required. If a patient is of childbearing potential the patient must agree to use effective contraception (see Appendix C for acceptable methods) during the study and for 120 days after the last dose of study drug. Non-childbearing potential is defined as (by other than medical reasons):
* ≥45 years of age and has not had menses for >2 years
* Amenorrheic for <2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation
* Post hysterectomy, oophorectomy or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 120 days after the last dose of study drug
* If male, agrees to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of study drug
* Life expectancy of greater than 3 months
* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Adequate bone-marrow, liver, and renal function as assessed by the following laboratory requirements within 4 weeks of starting treatment

  * Absolute neutrophil count >1,500 per uL
  * Hemoglobin > 9 g/dL
  * Platelets >100,000 per uL
  * Creatinine < 1.5 x ULN OR Creatinine clearance (CrCl) > 60 by Cockcroft-Gault Equation if Creatinine >1.5
  * AST and ALT < 2.5 x ULN (< 5 x ULN if documented liver metastases)
  * Total bilirubin <1.5 ULN OR direct bilirubin < ULN if total bilirubin > 1.5 x ULN
  * INR < 2.0
* Experienced resolution of toxic effect(s) of the most recent prior anti-cancer therapy to Grade <1 (except alopecia or neuropathy). If patient underwent major surgery or radiation therapy of >30 Gy, they must have recovered from the toxicity and/or complications from the intervention.

Exclusion Criteria

* History or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator, including, but not limited to:

  1. Myocardial infarction or arterial thromboembolic events within 6 months prior to screening or severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease, or a QTc interval > 470 msec.
  2. Uncontrolled hypertension or diabetes mellitus.
  3. Another known malignancy that is progressing or requires active treatment.
  4. Any prior history of other cancer within the prior 5 years with the exception of adequately treated basal cell carcinoma or cervical intraepithelial neoplasia [CIN]/cervical carcinoma in situ or melanoma in situ).
  5. Active infection requiring systemic therapy
  6. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Any contraindication to oral agents or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the investigator, would preclude adequate absorption.
* Allergy to benzamide, inactive components of entinostat, or any of the other administered therapies
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug.
* If female, is pregnant or breastfeeding.
* Known G6PD deficiency, severe psoriasis, porphyria, macular degeneration, or severe diabetic retinopathy due to greater potential HCQ toxicity
* Patients with pre-existing hypertension should be on a stable antihypertensive regimen and have a blood pressure ≤ 150/100 mmHg at the time of enrollment.
* Evidence or history of bleeding diathesis. Any hemorrhage or bleeding event of CTCAE grade 3 or higher within 4 weeks of start of study medication
* Non-healing wound, ulcer, or bone fracture
* Patients using warfarin are excluded. Patients using other oral or parenteral anticoagulation are not excluded provided they are on a stable dose of anticoagulant but must undergo more frequent platelet count monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Karasic TB, Brown TJ, Schneider C, Teitelbaum UR, Reiss KA, Mitchell TC, Massa RC, O'Hara MH, DiCicco L, Garcia-Marcano L, Amaravadi RK, O'Dwyer PJ. Phase I Trial of Regorafenib, Hydroxychloroquine, and Entinostat in Metastatic Colorectal Cancer. Oncologist. 2022 Sep 2;27(9):716-e689. doi: 10.1093/oncolo/oyac078. PMID 35552447

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: hydroxychloroquine: 600mg daily
  entinostat: 3mg weekly
  regorafenib: 160mg daily
- Dose Level 2: hydroxychloroquine: 600mg daily
  entinostat: 5mg weekly
  regorafenib: 160mg daily
- Dose Level 3: hydroxychloroquine: 1200mg daily
  entinostat: 5mg weekly
  regorafenib: 160mg daily
Period: Dose Level 1
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 6 | 0 | 0
Completed | 6 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Dose Level 2
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 0 | 7 | 0
Completed | 0 | 6 | 0
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Dose Level 3
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 0 | 0 | 7
Completed | 0 | 0 | 6
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: Regorafenib: 160mg daily 1-21 of 28 day cycle (with provisions to lower the starting dose to 80mg if toxicity is excessive)
  entinostat: 3mg weekly
  hydroxychloroquine: 600 daily
- Dose Level 2: Regorafenib: 160mg daily 1-21 of 28 day cycle (with provisions to lower the starting dose to 80mg if toxicity is excessive)
  entinostat: 5mg weekly
  hydroxychloroquine: 600 daily
- Dose Level 3: Regorafenib: 160mg daily 1-21 of 28 day cycle (with provisions to lower the starting dose to 80mg if toxicity is excessive)
  entinostat: 5mg weekly
  hydroxychloroquine: 1200mg daily
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 6 | 7 | 7 | 20
Age, Continuous [Median (Full Range); unit: years] | 65 [38 to 68] | 60 [41 to 74] | 69 [52 to 82] | 64.5 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 10
  Male | 3 | 4 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 7 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 5 | 7 | 6 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Hydroxychloroquine and Entinostat in Combination With Regorafenib
Description: Participants were evaluable for toxicity if they have taken one dose of HCQ and one dose of entinostat. To be considered for evaluability in a Phase I cohort in the absence of dose-limiting toxicity, patients should have completed > 85% of HCQ doses, and at least 3 of 4 entinostat doses. The MTD will be defined as a) the dose producing DLT in 1 out of 6 patients, or b) the dose level below the dose which produced DLT in ≥ 2 out of 3 patients, or in ≥ 2 out of 6 patients. DLTs will be defined by toxicity occurring during the first 4 weeks of this study.
Time Frame: 18 months
Measure: Number; unit: mg
Groups:
- All Participants: All participants who received at least 1 dose of hydroxychloroquine 1 dose of entinostat.
Arm/Group | All Participants
Number analyzed (Participants) | 20
mg
  Hydroxychloroquine Daily | 1200
  Entinostat weekly | 5

ADVERSE EVENTS:
Time Frame: up to 18 months
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/7 | 6/7
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=7) | Dose Level 3 (N=7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombolicevent (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Rectal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=6) | Dose Level 2 (N=7) | Dose Level 3 (N=7)
Anemia (Blood and lymphatic system disorders) | 1 | 3 | 3
Bloating (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis Oral (Gastrointestinal disorders) | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Fatigue (General disorders) | 3 | 3 | 4
Fever (General disorders) | 1 | 0 | 0
Gait Disturbance (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Mucosal Infection (Infections and infestations) | 1 | 0 | 1
Papulopustular Rash (Infections and infestations) | 1 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 1
Weight loss (Investigations) | 3 | 3 | 6
White Blood Cell Decreased (Investigations) | 1 | 3 | 3
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Platelet Count Decreased (Investigations) | 2 | 2 | 4
Alkaline Phosphate Increased (Investigations) | 3 | 1 | 5
Aspartate Aminotransferase Increased (Investigations) | 2 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 0
Thyroid Stimulating Hormone Increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 4 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Urinary Frequency (Renal and urinary disorders) | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Palmer-plantar erthrodysesthesia (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Puritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03215264/Prot_SAP_000.pdf